CLINICAL TRIAL: NCT01520909
Title: A Two Part, Double-blind, Randomized, Placebo-controlled and Open-label Study to Investigate the Efficacy, Safety and Tolerability of Eltrombopag, a Thrombopoietin Receptor Agonist, in Pediatric Patients With Previously Treated Chronic Immune (Idiopathic) Thrombocytopenic Purpura (ITP). PETIT2: Eltrombopag in PEdiatric Patients With Thrombocytopenia From ITP
Brief Title: Study of a New Medication for Childhood Chronic Immune Thrombocytopenia (ITP), a Blood Disorder of Low Platelet Counts That Can Lead to Bruising Easily, Bleeding Gums, and/or Bleeding Inside the Body.
Acronym: PETIT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115450; 2011-002184-17 (EudraCT Number)
Record Dates: First submitted 2011-12-21; First posted 2012-01-30 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-02

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: immune thrombocytopenic purpura; pediatrics; chronic ITP; idiopathic thrombocytopenic purpura; eltrombopag; Chronic Immune Thrombocytopenia; platelet disorder; thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Blood Platelet Disorders; Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Eltrombopag plus standard of care (Experimental): Part 1, double-blind treatment group
  Interventions: Drug: Eltrombopag
- Placebo plus standard of care (Placebo Comparator): Part 1, double-blind treatment group
  Interventions: Drug: Placebo
- Eltrombopag plus standard of care (Part 2 open-label) (Experimental): Part 2, open-label
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Thrombopoietin receptor agonist
  Arms: Eltrombopag plus standard of care; Eltrombopag plus standard of care (Part 2 open-label)
Drug: Placebo — Placebo with no active pharmaceutical ingredient
  Arms: Placebo plus standard of care

SUMMARY:
The purpose of this study is to investigate the efficacy, safety and tolerability of eltrombopag in children with previously treated chronic immune thrombocytopenia who are between 1 and 17 years of age. This is a 2 part study. In part 1, patients will be randomized to receive either eltrombopag or placebo for 13 weeks. All patients who complete part 1 will enter part 2. In part 2, all patients will receive 24 weeks of eltrombopag.

DETAILED DESCRIPTION:
This is a two part, double-blind, randomized, placebo-controlled and open-label Phase III study to investigate the efficacy, safety and tolerability of eltrombopag in pediatric patients with previously treated chronic ITP. In Part 1, patients will be randomized to receive eltrombopag or placebo in a 13-week double-blind, placebo-controlled treatment period. After completing Part 1, patients will begin Part 2, in which they will receive eltrombopag in an open-label manner during a 24-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained from the patient's guardian and accompanying informed assent from the patient (for children over 6 years old)
* Patients must be between 1 year and <18 years of age at Day 1
* Patients will have a confirmed diagnosis of chronic ITP for at least 1 year, at screening, according to the guidelines published in the International Working Group Report
* A peripheral blood smear or bone marrow examination will support the diagnosis of ITP with no evidence of other causes of thrombocytopenia.
* Patients must be refractory or have relapsed after at least one prior ITP therapy, or patients must be unable, for a medical reason, to continue other ITP treatments.
* Patients must have a Day 1 (or within 48 hours prior) platelet count <30 Gi/L.
* Previous therapy for ITP with immunoglobulins (IVIg and anti-D) must have been completed at least 2 weeks prior to Day 1, or these therapies must have been completed at least 1 week prior to Day 1 and have been clearly ineffective.
* Previous treatment for ITP with splenectomy, rituximab and cyclophosphamide must have been completed at least 4 weeks prior to Day 1.
* Patients treated with concomitant ITP medication (e.g. corticosteroids or azathioprine) must be receiving a dose that has been stable for at least 4 weeks prior to Day 1.
* Patients must have a complete blood count (CBC) not suggestive of another hematological disorder.
* Patients must have the following laboratory results:
* prothrombin time international normalized ratio (INR) and activated partial thromboplastin time (aPTT) within 80 to 120% of the normal range.
* clinical chemistries that do NOT exceed the upper limit of normal reference range by more than 20% for the following: creatinine, ALT, AST, total bilirubin, and alkaline phosphatase.
* total albumin that is not below the lower limit of normal by more than 10%.
* Female patients of child-bearing potential (after menarche) must:
* have a negative pregnancy test within 24 hours of first dose of study treatment,
* agree and be able to provide a blood or urine specimen for pregnancy testing during the study,
* agree to use effective contraception during the study and for 28 days following the last dose of study treatment, and not be lactating.
* Male patients with a female partner of childbearing potential must agree to use effective contraception from 2 weeks prior to administration of the first dose of study treatment until 3 months after the last dose of study treatment.
* In France, a patient will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Patients with any clinically relevant abnormality, other than ITP, identified on the screening examination or any other medical condition or circumstance, which in the opinion of the investigator makes the patient unsuitable for participation in the study or suggests another primary diagnosis (e.g. Thrombocytopenia is secondary to another disease).
* Patients with concurrent or past malignant disease, including myeloproliferative disorder.
* Patients expected not to be suitable for continuation of their current therapy for at least 13 additional weeks.
* Patients with a history of platelet agglutination abnormality that prevents reliable measurement of platelet counts.
* Patients with a diagnosis of secondary immune thrombocytopenia, including those with laboratory or clinical evidence of HIV infection, anti-phospholipid antibody syndrome, chronic hepatitis B infection, hepatitis c virus infection, or any evidence of active hepatitis at the time of subject screening.
* Patients with Evans syndrome (autoimmune thrombocytopenia and autoimmune hemolysis).
* Patients with known inherited thrombocytopenia (e.g. MYH9 disorders).
* Patients treated with any medication that affects platelet function (including but not limited to aspirin, clopidogrel and/or NSAIDS) or anti-coagulants for >3 consecutive days within 2 weeks of Day 1.
* Patients who have received treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding Day 1.
* Patients who have previously received eltrombopag or any other thrombopoietin receptor agonist.
* Any patient considered to be a child in care, defined as one who has been placed under the control or protection of an agency, organization, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation. This can include a child cared for by foster parents or living in a care home or institution, provided that the arrangement falls within the definition above. The definition of a child in care does not include a child who is adopted or who has an appointed legal guardian.
* Patients who have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to eltrombopag or excipients that contraindicates their participation.
* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions that could interfere with the patient's safety or compliance to the study procedures.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (48):
- United States (4):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Salt Lake City, Utah
- GSK Investigational Site, Capital Federal, Buenos Aires, Argentina
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Prague
- Germany (3):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Berlin, State of Berlin
- Hong Kong (2):
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shatin
- Israel (6):
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Rehovot
  - GSK Investigational Site, Tel Aviv
- Italy (4):
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Monza, Lombardy
  - GSK Investigational Site, Turin, Piedmont
- Poland (4):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
- Russia (3):
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- Spain (6):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Murcia (El Palmar)
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Valencia
- Taiwan (2):
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taoyuan District
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Songkhla
- United Kingdom (6):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Romford
  - GSK Investigational Site, Sheffield

REFERENCES:
- [Derived] Wire MB, Li X, Zhang J, Sallas W, Aslanis V, Ouatas T. Modeling and Simulation Support Eltrombopag Dosing in Pediatric Patients With Immune Thrombocytopenia. Clin Pharmacol Ther. 2018 Dec;104(6):1199-1207. doi: 10.1002/cpt.1066. Epub 2018 Apr 17. PMID 29536526
- [Derived] Grainger JD, Locatelli F, Chotsampancharoen T, Donyush E, Pongtanakul B, Komvilaisak P, Sosothikul D, Drelichman G, Sirachainan N, Holzhauer S, Lebedev V, Lemons R, Pospisilova D, Ramenghi U, Bussel JB, Bakshi KK, Iyengar M, Chan GW, Chagin KD, Theodore D, Marcello LM, Bailey CK. Eltrombopag for children with chronic immune thrombocytopenia (PETIT2): a randomised, multicentre, placebo-controlled trial. Lancet. 2015 Oct 24;386(10004):1649-58. doi: 10.1016/S0140-6736(15)61107-2. Epub 2015 Jul 28. PMID 26231455

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric participants meeting eligibility criteria were enrolled into 3 cohorts depending upon age. Cohort 1 enrolled participants who were between 12 and 17 years old, Cohort 2 enrolled participants who were between 6 and 11 years old, and Cohort 3 enrolled participants who were between 1 and 5 years old.
Pre-assignment Details: This study was comprised of a 13-week Double-Blind (DB), randomized Treatment Period (Part 1), followed by a 24-week Open-Label (OL) eltrombopag-only period (Part 2). After completion of Part 2, participants completed a 24- to 28-week Follow-up period, including an ophthalmic examination 24 weeks after the last dose of study treatment.
Groups:
- Part 1 (Randomized Period)-Placebo: In Part 1, participants aged between 6 and 17 years with a body weight <27 kilograms (kg) received placebo 37.5 milligrams (mg) once daily (QD), and those with a body weight >=27 kg received placebo 50 mg QD. Participants of East Asian ancestry received a starting dose of placebo 25 mg QD. Participants aged between 1 and 5 years received placebo 1.2 milligrams per kilogram (mg/kg) QD; participants of East Asian ancestry received a starting dose of placebo 0.8 milligrams per kilograms per day (mg/kg/day). Standard of care treatments were allowed during the study, and were prescribed based on the investigator's discretion.
- Part 1 (Randomized Period)-Eltrombopag: In Part 1, participants aged between 6 and 17 years with a body weight <27 kg received eltrombopag 37.5 mg QD, and those with a body weight >=27 kg received eltrombopag 50 mg QD. Participants of East Asian ancestry received a starting dose of eltrombopag 25 mg QD. Participants aged between 1 and 5 years received eltrombopag 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of eltrombopag 0.8 mg/kg/day. Participants continued on the same dose of eltrombopag in Part 2 unless adjustments were warranted according to the dosing guidelines. Standard of care treatments were allowed during the study, and were prescribed based on the investigator's discretion.
- Part 2 (Open-Label Period) Eltrombopag: All participants receiving placebo in Part 1 received eltrombopag in Part 2 following starting dose guidelines for Part 1. Participants aged between 6 and 17 years with a body weight <27 kg received eltrombopag 37.5 mg QD, and those with a body weight >=27 kg received eltrombopag 50 mg QD. Participants of East Asian ancestry received a starting dose of eltrombopag 25 mg QD. Participants aged between 1 and 5 years received eltrombopag 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of eltrombopag 0.8 mg/kg/day. Participants receiving eltrombopag in Part 1 continued on the same dose of eltrombopag in Part 2 unless adjustments were warranted according to the dosing guidelines. Standard of care treatments were allowed during the study, and were prescribed based on the investigator's discretion.
Period: Part 1 (Randomized Period)
Arm/Group | Part 1 (Randomized Period)-Placebo | Part 1 (Randomized Period)-Eltrombopag | Part 2 (Open-Label Period) Eltrombopag
Started | 29 | 63 | 0
Completed | 28 | 61 | 0
Not Completed | 1 | 2 | 0
Not completed — Adverse Event | 1 | 2 | 0
Period: Part 2 (Open-Label Period)-Eltrombopag
Arm/Group | Part 1 (Randomized Period)-Placebo | Part 1 (Randomized Period)-Eltrombopag | Part 2 (Open-Label Period) Eltrombopag
Started | 0 | 0 | 87 (Two participants that completed Part 1 did not start Part 2 because of lack of efficacy.)
Completed | 0 | 0 | 80
Not Completed | 0 | 0 | 7
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Withdrawal by parent or guardian | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: In Part 1, participants aged between 6 and 17 years with a body weight <27 kg received placebo 37.5 mg QD, and those with a body weight >=27 kg received placebo 50 mg QD. Participants of East Asian ancestry received a starting dose of placebo 25 mg QD. Participants aged between 1 and 5 years received placebo 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of placebo 0.8 mg/kg/day. In Part 2, participants received eltrombopag. Participants aged between 6 and 17 years with a body weight <27 kg received eltrombopag 37.5 mg QD, and those with a body weight >=27 kg received eltrombopag 50 mg QD. Participants of East Asian ancestry received a starting dose of eltrombopag 25 mg QD. Participants aged between 1 and 5 years received eltrombopag 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of eltrombopag 0.8 mg/kg/day.
- Eltrombopag: In Part 1, participants aged between 6 and 17 years with a body weight <27 kg received eltrombopag 37.5 mg QD, and those with a body weight >=27 kg received eltrombopag 50 mg QD. Participants of East Asian ancestry received a starting dose of eltrombopag 25 mg QD. Participants aged between 1 and 5 years received eltrombopag 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of eltrombopag 0.8 mg/kg/day. Participants continued on the same dose of eltrombopag in Part 2 unless adjustments were warranted according to the dosing guidelines.
- Total: Total of all reporting groups
Arm/Group | Placebo | Eltrombopag | Total
Number analyzed (Participants) | 29 | 63 | 92
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.8 (4.00) | 9.4 (4.43) | 9.6 (4.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 30 | 44
  Male | 15 | 33 | 48
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 0 | 1 | 1
  Central/South Asian Heritage | 0 | 1 | 1
  Japanese/East Asian/South East Asian Heritage | 10 | 20 | 30
  Arabic/North African Heritage | 1 | 2 | 3
  White/Caucasian/European Heritage | 18 | 38 | 56
  Mixed Race | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving a Platelet Count >=50 Giga Cells Per Liter (Gi/L) for at Least 6 Out of 8 Weeks, Between Weeks 5 and 12 of Part 1
Description: Participants who achieved a platelet count >=50 Gi/L for at least 6 out of 8 weeks, between Weeks 5 and 12 of Part 1, were reported.
Time Frame: From Week 5 up to Week 12 of Part 1
Population: Intent-to-Treat (ITT) Population: all randomized participants. The ITT Population was the primary population used for assessing efficacy.
Measure: Number; unit: Participants
Groups:
- Part 1 (Randomized Period)- Placebo: In Part 1, participants aged between 6 and 17 years with a body weight <27 kilograms (kg) received placebo 37.5 milligrams (mg) once daily (QD), and those with a body weight >=27 kg received placebo 50 mg QD. Participants of East Asian ancestry received a starting dose of placebo 25 mg QD. Participants aged between 1 and 5 years received placebo 1.2 milligrams per kilogram (mg/kg) QD; participants of East Asian ancestry received a starting dose of placebo 0.8 milligrams per kilograms per day (mg/kg/day).
- Part 1 (Randomized Period)-Eltrombopag: In Part 1, participants aged between 6 and 17 years with a body weight <27 kg received eltrombopag 37.5 mg QD, and those with a body weight >=27 kg received eltrombopag 50 mg QD. Participants of East Asian ancestry received a starting dose of eltrombopag 25 mg QD. Participants aged between 1 and 5 years received eltrombopag 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of eltrombopag 0.8 mg/kg/day.
Arm/Group | Part 1 (Randomized Period)- Placebo | Part 1 (Randomized Period)-Eltrombopag
Number analyzed (Participants) | 29 | 63
Participants | 1 | 25
Statistical Analysis 1: Comparison: Part 1 (Randomized Period)- Placebo vs Part 1 (Randomized Period)-Eltrombopag; Indicated significance at the 5% (two-sided) level of significance; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; The proportion of participants achieving platelet counts >=50 Gi/L for those participants receiving eltrombopag versus placebo was compared; Odds Ratio (OR) = 17.96, 95% CI 2-sided [2.29 to 140.93]

2. Secondary Outcome: Percentage of Responders
Description: Percentage of participants who responded (defined as platelet count >= 50 Gi/L in absence of rescue) at least once up to week 12 of Part 1 (Odds of achieving a platelet count >=50 Gi/L during the first 12 weeks of Part 1)
Time Frame: From Week 1 up to Week 12 of Part 1
Population: ITT Population
Measure: Number; unit: Percentage of participants
Groups:
- Part 1 (Randomized Period)-Placebo: In Part 1, participants aged between 6 and 17 years with a body weight <27 kg received placebo 37.5 mg QD, and those with a body weight >=27 kg received placebo 50 mg QD. Participants of East Asian ancestry received a starting dose of placebo 25 mg QD. Participants aged between 1 and 5 years received placebo 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of placebo 0.8 mg/kg/day.
- Part 1 (Randomized Period) - Eltrombopag: In Part 1, participants aged between 6 and 17 years with a body weight <27 kg received eltrombopag 37.5 mg QD, and those with a body weight >=27 kg received eltrombopag 50 mg QD. Participants of East Asian ancestry received a starting dose of eltrombopag 25 mg QD. Participants aged between 1 and 5 years received eltrombopag 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of eltrombopag 0.8 mg/kg/day.
Arm/Group | Part 1 (Randomized Period)-Placebo | Part 1 (Randomized Period) - Eltrombopag
Number analyzed (Participants) | 29 | 63
Percentage of participants
  Week 1 | 0 | 15.9
  Week 2 | 3.4 | 23.8
  Week 3 | 0 | 31.7
  Week 4 | 6.9 | 36.5
  Week 5 | 6.9 | 47.6
  Week 6 | 6.9 | 38.1
  Week 7 | 10.3 | 44.4
  Week 8 | 3.4 | 44.4
  Week 9 | 3.4 | 42.9
  Week 10 | 3.4 | 52.4
  Week 11 | 6.9 | 49.2
  Week 12 | 3.4 | 58.7
Statistical Analysis 1: Comparison: Part 1 (Randomized Period)-Placebo vs Part 1 (Randomized Period) - Eltrombopag; Test type: Superiority or Other; p < 0.001, Repeated measures model for binary data; Repeated measures model for binary data using Generalized linear mixed model; Odds Ratio (OR) = 25.33, 95% CI 2-sided [8.15 to 78.73]

3. Secondary Outcome: Number of Participants Achieving a Platelet Count >=50 Gi/L at Any Time During the First 12 Weeks of Part 1
Description: Participants who achieved a platelet count >=50 Gi/L at any time during the first 12 weeks of Part 1 were reported.
Time Frame: From Baseline up to Week 12 of Part 1
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Part 1 (Randomized Period)-Placebo | Part 1 (Randomized Period) - Eltrombopag
Number analyzed (Participants) | 29 | 63
Participants | 6 | 47

4. Secondary Outcome: Number of Participants Achieving a Platelet Count >=50 Gi/L at Any Time During the First 6 Weeks of Part 1
Description: Participants who achieved a platelet count >=50 Gi/L at any time during the first 6 weeks of Part 1 were reported.
Time Frame: From Baseline up to Week 6 of Part 1
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Part 1 (Randomized Period)-Placebo | Part 1 (Randomized Period)-Eltrombopag
Number analyzed (Participants) | 29 | 63
Participants | 5 | 39

5. Secondary Outcome: Weighted Mean Platelet Count
Description: The weighted mean platelet count is defined as "the area under the platelet-time curve divided by the duration of the study (12 weeks)". Weighted mean platelet counts from baseline to week 12 of the randomized period was compared between placebo and eltrombopag using an analysis of covariance model (ANCOVA) adjusting for baseline platelet count and age cohort. For each subject the area between two adjacent visits with platelet counts was calculated. The area was calculated for all pairs of adjacent visits starting at Day 1 of randomized period and then the total sum of all the areas was divided by the total duration of time during the randomized period. For each subject, this method calculates an 'average' platelet count and it allows the possibility that subjects may have had different number of assessments during different times relative to baseline.
Time Frame: Baseline and Week 12 of Part 1
Population: ITT Population. Only those participants with a value at Baseline and post-Baseline were analyzed.
Measure: Mean (Standard Deviation); unit: Gi/L
Arm/Group | Part 1 (Randomized Period)-Placebo | Part 1 (Randomized Period) - Eltrombopag
Number analyzed (Participants) | 29 | 62
Gi/L
  Baseline | 14.2 (8.01) | 14.0 (8.09)
  Week 12 | 23.7 (19.56) | 63.9 (46.68)

6. Secondary Outcome: Maximum Duration for Which a Participant Continuously Maintained a Platelet Count of >=50 Gi/L During the First 12 Weeks of Part 1
Description: The maximum duration for which a participant continuously maintained a platelet count >=50 Gi/L was calculated and summarized for the first 12 weeks of Part 1. Participants with non-weekly assessments were assumed to have maintained a positive response for each week between two assessments that had positive responses. If a participant achieved a positive response at an assessment and then achieved a negative response at the next assessment, then it was assumed that the participant had achieved a positive response for one day.
Time Frame: From Baseline up to Week 12 of Part 1
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Part 1 (Randomized Period)-Placebo | Part 1 (Randomized Period) - Eltrombopag
Number analyzed (Participants) | 29 | 63
Weeks | 0.4 (1.50) | 3.3 (3.13)

7. Secondary Outcome: Number of Participants Who Required a Protocol-defined Rescue Treatment During Part 1
Description: Rescue treatment is defined as either a new immune (idiopathic) thrombocytopenic purpura (ITP) medication, an increase in the dose of a concomitant ITP medication from Baseline, a platelet transfusion, or a splenectomy.
Time Frame: From Baseline up to Week 12 of Part 1
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Part 1 (Randomized Period)-Placebo | Part 1 (Randomized Period) - Eltrombopag
Number analyzed (Participants) | 29 | 63
Participants | 7 | 12

8. Secondary Outcome: Number of Participants With Any Bleeding and Significant Bleeding as Assessed Using the World Health Organization (WHO) Bleeding Scale During Part 1
Description: The WHO Bleeding Scale is a measure of bleeding severity with the following grades: Grade 0=no bleeding; Grade 1=petechiae; Grade 2=mild blood loss; Grade 3=gross bleeding; Grade 4=debilitating blood loss. The WHO grades were dichotomized into the following categories: no bleeding=Grade 0; any bleeding=Grades 1 to 4; no clinically significant bleeding=Grades 0 to 1; clinically significant bleeding=Grades 2 to 4. Baseline was defined as the Day 1 assessment or the latest possible screening assessment.
Time Frame: From Baseline through Follow-up of Part 1
Population: ITT Population. Only those participants that did not enroll in Part 2 were analyzed during the follow-up visits. Only those participants available at the specified time points were analyzed (represented by n=X,X in the category titles).
Measure: Number; unit: Participants
Groups:
- Part 1 (Randomized Period) -Eltrombopag: In Part 1, participants aged between 6 and 17 years with a body weight <27 kg received eltrombopag 37.5 mg QD, and those with a body weight >=27 kg received eltrombopag 50 mg QD. Participants of East Asian ancestry received a starting dose of eltrombopag 25 mg QD. Participants aged between 1 and 5 years received eltrombopag 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of eltrombopag 0.8 mg/kg/day.
Arm/Group | Part 1 (Randomized Period)-Placebo | Part 1 (Randomized Period) -Eltrombopag
Number analyzed (Participants) | 29 | 63
Participants
  Baseline, Any bleeding n=29,63 | 20 | 45
  Baseline, Significant bleeding n=29,63 | 6 | 16
  Week 1, Any bleeding n=29,63 | 19 | 41
  Week 1, Significant bleeding n=29,63 | 3 | 8
  Week 2, Any bleeding n=29,63 | 19 | 33
  Week 2, Significant bleeding n=29,63 | 6 | 6
  Week 3, Any bleeding n=28,62 | 18 | 32
  Week 3, Significant bleeding n=28,62 | 3 | 7
  Week 4, Any bleeding n=29, 62 | 20 | 27
  Week 4, Significant bleeding n=29, 62 | 4 | 4
  Week 5, Any bleeding n=27, 62 | 18 | 22
  Week 5, Significant bleeding n=27, 62 | 2 | 5
  Week 6, Any bleeding n=28, 62 | 17 | 24
  Week 6, Significant bleeding n=28, 62 | 0 | 5
  Week 7, Any bleeding n=28, 63 | 14 | 20
  Week 7, Significant bleeding n=28, 63 | 1 | 1
  Week 8, Any bleeding n=28, 63 | 17 | 24
  Week 8,Significant bleeding n=28, 63 | 1 | 4
  Week 9, Any bleeding n=27, 61 | 18 | 24
  Week 9, Significant bleeding n=27, 61 | 3 | 4
  Week 10, Any bleeding n=28, 62 | 17 | 20
  Week 10, Significant bleeding n=28, 62 | 2 | 4
  Week 11, Any bleeding n=28, 61 | 16 | 26
  Week 11, Significant bleeding n=28, 61 | 3 | 8
  Week 12, Any bleeding n=28, 61 | 16 | 23
  Week 12, Significant bleeding n=28, 61 | 2 | 3
  Follow-up Week 1, Any bleeding n=0,2 | 0 | 1
  Follow-up Week 1, Significant bleeding n=0,2 | 0 | 0
  Follow-up Week 2, Any bleeding n=0,2 | 0 | 1
  Follow-up Week 2, Significant bleeding n=0,2 | 0 | 0
  Follow-up Week 3, Any bleeding n=0,3 | 0 | 2
  Follow-up Week 3, Significant bleeding n=0,3 | 0 | 1
  Follow-up Week 4, Any bleeding n=0,1 | 0 | 1
  Follow-up Week 4, Significant bleeding n=0,1 | 0 | 1
  Any follow-up Week, Any bleeding n=0,3 | 0 | 2
  Any Follow-up Week, Significant bleeding n=0,3 | 0 | 1

9. Secondary Outcome: Number of Participants Who Achieved a Platelet Count >=50 Gi/L at Any Time During Part 2
Description: Participants who achieved a platelet count >=50 Gi/L at any time during Part 2 (up to Week 24) were reported.
Time Frame: From Baseline up to Week 24 of Part 2
Population: ITT Population. Only those participants who entered into Part 2 (Open-label eltrombopag-only phase) were analyzed.
Measure: Number; unit: Participants
Groups:
- Part 2 (Open-Label Period) - Eltrombopag: Participants who received eltrombopag in Part 1 continued on the same dose in Part 2 unless adjustments were warranted according to the dosing guidelines. Participants who received placebo in Part 1 received Eltrombopag as per age criteria as follows: aged between 6 and 17 years with a body weight <27 kg received eltrombopag 37.5 mg QD, and those with a body weight >=27 kg received eltrombopag 50 mg QD. Participants of East Asian ancestry received a starting dose of eltrombopag 25 mg QD. Participants aged between 1 and 5 years received eltrombopag 1.2 mg/kg QD and; participants of East Asian ancestry received a starting dose of eltrombopag 0.8 mg/kg/day.
Arm/Group | Part 2 (Open-Label Period) - Eltrombopag
Number analyzed (Participants) | 87
Participants | 70

10. Secondary Outcome: Number of Weeks in Which Participants Achieved a Platelet Count >=50 Gi/L, Between Weeks 4 and 24 of Part 2
Description: Platelet response was analyzed after Week 4 for the eltrombopag-only period to allow participants who had been randomized to placebo in the Randomized Period time to escalate to their optimal dose of eltrombopag. Participants with non-weekly assessments were assumed to have maintained a positive response for each week between two assessments that had positive responses. If the participant achieved a positive response at an assessment and then achieved a negative response at the next assessment, then it was assumed that the participant had achieved a positive response for one day.
Time Frame: From Week 4 up to Week 24 of Part 2
Population: ITT Population. Only those participants who entered into Part 2 (Open-label eltrombopag-only phase) were analyzed.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Part 2 (Open-Label Period) - Eltrombopag
Number analyzed (Participants) | 87
Weeks | 10 (7.67)

11. Secondary Outcome: Maximum Duration for Which a Participant Continuously Maintained a Platelet Count of >=50 Gi/L During Part 2
Description: The maximum duration for which a participant continuously maintained a platelet count of >=50 Gi/L was calculated and summarized for the 24 weeks of eltrombopag dosing (Part 2). Participants with non-weekly assessments were assumed to have maintained a positive response for each week between two assessments that had positive responses. If the participant achieved a positive response at an assessment and then achieved a negative response at the next assessment, then it was assumed that the participant had achieved a positive response for one day.
Time Frame: From Baseline up to Week 24 of Part 2
Population: ITT Population. Only those participants who entered into Part 2 (Open-label eltrombopag-only phase) were analyzed.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Part 2 (Open-Label Period) - Eltrombopag
Number analyzed (Participants) | 87
Weeks | 8.6 (7.84)

12. Secondary Outcome: Number of Participants Who Reduced or Discontinued Baseline Concomitant ITP Medications During Part 2 Without Requiring Subsequent Rescue Therapy
Description: Participants who discontinued or had a sustained reduction of a baseline immune (idiopathic) thrombocytopenic purpura (ITP) medication during the 24 weeks of Part 2 (Open-Label Period) and without requiring subsequent rescue therapy. For participants randomized to placebo in Part 1, Baseline is defined as Week 13 of Part 1. For participants randomized to eltrombopag in Part 1, Baseline is defined as Day 1 of Part 1. A sustained reduction was defined as a reduction for 4 weeks or more.
Time Frame: From Baseline up to Week 24 of Part 2
Population: ITT Population. Only those participants who entered into Part 2 (Open-label eltrombopag-only phase) and taking an ITP medication at Baseline were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 2 (Open-Label Period) - Eltrombopag
Number analyzed (Participants) | 15
Participants | 8

13. Secondary Outcome: Number of Participants Who Required a Protocol-defined Rescue Treatment During Part 2
Description: Rescue treatment was defined as either a new immune (idiopathic) thrombocytopenic purpura (ITP) medication, an increase in the dose of a concomitant ITP medication from Baseline, a platelet transfusion, or a splenectomy.
Time Frame: From Baseline up to Week 24 of Part 2
Population: ITT Population. Only those participants who entered into Part 2 (Open-label eltrombopag-only phase) were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 2 (Open-Label Period) - Eltrombopag
Number analyzed (Participants) | 87
Participants | 11

14. Secondary Outcome: Number of Participants With Any Bleeding and Significant Bleeding as Assessed Using the WHO Bleeding Scale During Part 2
Description: The WHO Bleeding Scale is a measure of bleeding severity with the following grades: Grade 0 = no bleeding, Grade 1 = petechiae, Grade 2 = mild blood loss, Grade 3 = gross bleeding and Grade 4 = debilitating blood loss. The WHO Grades were dichotomized into the following categories: no bleeding = Grade 0; any bleeding = Grade 1 to 4; no clinically significant bleeding = Grade 0 to 1; clinically significant bleeding = Grade 2 to 4.
Time Frame: From Baseline of Part 2 through Follow-up
Population: ITT Population. Only those participants who entered into Part 2 open-label Eltrombopag only phase were analyzed. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Number; unit: Participants
Arm/Group | Part 2 (Open-Label Period) - Eltrombopag
Number analyzed (Participants) | 87
Participants
  Baseline, Any bleeding n=87 | 55
  Baseline, Significant bleeding n=87 | 17
  Week 1, Any bleeding n=86 | 29
  Week 1, Significant bleeding n=86 | 3
  Week 2, Any bleeding n=85 | 22
  Week 2, Significant bleeding n=85 | 2
  Week 3, Any bleeding n=86 | 20
  Week 3, Significant bleeding n=86 | 1
  Week 4, Any bleeding n=68 | 20
  Week 4, Significant bleeding n=68 | 4
  Week 5, Any bleeding n=61 | 21
  Week 5, Significant bleeding n=61 | 4
  Week 6, Any bleeding n=55 | 17
  Week 6, Significant bleeding n=55 | 3
  Week 7, Any bleeding n=52 | 14
  Week 7, Significant bleeding n=52 | 1
  Week 8, Any bleeding n=52 | 17
  Week 8, Significant bleeding n=52 | 4
  Week 9, Any bleeding n=45 | 11
  Week 9, Significant bleeding n=45 | 1
  Week 10, Any bleeding n=42 | 8
  Week 10, Significant bleeding n=42 | 2
  Week 11, Any bleeding n=40 | 12
  Week 11, Significant bleeding n=40 | 3
  Week 12, Any bleeding n=63 | 15
  Week 12, Significant bleeding n=63 | 5
  Week 13, Any bleeding n=30 | 9
  Week 13, Significant bleeding n=30 | 2
  Week 14, Any bleeding n=38 | 9
  Week 14, Significant bleeding n=38 | 2
  Week 15, Any bleeding n=43 | 10
  Week 15, Significant bleeding n=43 | 2
  Week 16, Any bleeding n=47 | 11
  Week 16, Significant bleeding n=47 | 4
  Week 17, Any bleeding n=37 | 10
  Week 17, Significant bleeding n=37 | 2
  Week 18, Any bleeding n=33 | 8
  Week 18, Significant bleeding n=33 | 1
  Week 19, Any bleeding n=44 | 15
  Week 19, Significant bleeding n=44 | 2
  Week 20, Any bleeding n=39 | 7
  Week 20, Significant bleeding n=39 | 2
  Week 21, Any bleeding n=41 | 10
  Week 21, Significant bleeding n=41 | 2
  Week 22, Any bleeding n=34 | 7
  Week 22, Significant bleeding n=34 | 3
  Week 23, Any bleeding n=36 | 15
  Week 23, Significant bleeding n=36 | 2
  Week 24, Any bleeding n=79 | 19
  Week 24, Significant bleeding n=79 | 5
  Follow-up Week 1, Any bleeding n=29 | 8
  Follow-up Week 1, Significant bleeding n=29 | 2
  Follow-up Week 2, Any bleeding n=37 | 25
  Follow-up Week 2, Significant bleeding n=37 | 5
  Follow-up Week 3, Any bleeding n=40 | 17
  Follow-up Week 3, Significant bleeding n=40 | 5
  Follow-up Week 4, Any bleeding n=70 | 23
  Follow-up Week 4, Significant bleeding n=70 | 3
  Any follow-up Week, Any bleeding n=77 | 38
  Any Follow-up Week, Significant bleeding n=77 | 8

15. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE) During Part 1
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, or is a congenital anomaly or birth defect. Medical or scientific judgment should be exercised in other situations.
Time Frame: From Day 1 of Treatment up to Week 13 of Part 1+ 1 day
Population: Safety Population: all participants who received at least one dose of the investigational product
Measure: Number; unit: Participants
Groups:
- Part 1 (Randmoized Period) -Placebo: In Part 1, participants aged between 6 and 17 years with a body weight <27 kg received placebo 37.5 mg QD, and those with a body weight >=27 kg received placebo 50 mg QD. Participants of East Asian ancestry received a starting dose of placebo 25 mg QD. Participants aged between 1 and 5 years received placebo 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of placebo 0.8 mg/kg/day.
Arm/Group | Part 1 (Randmoized Period) -Placebo | Part 1 (Randomized Period) - Eltrombopag
Number analyzed (Participants) | 29 | 63
Participants
  Any AE | 21 | 51
  Any SAE | 4 | 5

16. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE) During Part 2
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death, is life threatening; requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, or is a congenital anomaly or birth defect. Medical or scientific judgment should be exercised in other situations.
Time Frame: From Day 1 of Part 2 up to Week 24 of Part 2 + 1 day
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part 2 (Open-Label Period) - Eltrombopag
Number analyzed (Participants) | 87
Participants
  Any AE | 69
  Any SAE | 9

17. Secondary Outcome: Number of Participants With the Indicated Maximum Toxicity Grade for the Indicated Clinical Chemistry Parameters at Any Time Post-Baseline During Part 1
Description: Clinical chemistry parameters were summarized according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0: Grade 0 (G0), none; Grade 1 (G1), mild; Grade 2 (G2), moderate; Grade 3 (G3), severe; Grade 4 (G4), life-threatening or disabling. Clinical chemistry parameters included: aspartate amino transferase (AST), alkaline phosphatase (ALP), total bilirubin, albumin, alanine amino transferase (ALT), prothrombin international normalized ratio (PT INR), activated partial thromboplastin time (APTT), and creatinine. The Baseline value is defined as the value taken at Day 1 or, if missing, the latest non-missing Screening value. For serum creatinine, due to the variations in creatinine, the average of the Screening and the Day 1 values will be used as Baseline. The maximum post-Baseline toxicity grade includes any scheduled or unscheduled post-Baseline assessment during Part 1.
Time Frame: From Baseline up to Week 13 of Part 1
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X,X in the category titles).
Measure: Number; unit: Participants
Groups:
- Part 1 (Randmoized Period)-Placebo: In Part 1, participants aged between 6 and 17 years with a body weight <27 kg received placebo 37.5 mg QD, and those with a body weight >=27 kg received placebo 50 mg QD. Participants of East Asian ancestry received a starting dose of placebo 25 mg QD. Participants aged between 1 and 5 years received placebo 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of placebo 0.8 mg/kg/day.
Arm/Group | Part 1 (Randmoized Period)-Placebo | Part 1 (Randomized Period) - Eltrombopag
Number analyzed (Participants) | 29 | 63
Participants
  AST, G0, n=29, 63 | 26 | 50
  AST, G1, n=29, 63 | 3 | 12
  AST, G2, n=29, 63 | 0 | 1
  AST, G3, n=29, 63 | 0 | 0
  AST, G4, n=29, 63 | 0 | 0
  ALT, G0, n=29, 63 | 27 | 52
  ALT, G1, n=29, 63 | 2 | 6
  ALT, G2, n=29, 63 | 0 | 3
  ALT, G3, n=29, 63 | 0 | 2
  ALT, G4, n=29, 63 | 0 | 0
  Total Bilirubin, G0, n=29, 63 | 29 | 60
  Total Bilirubin, G1, n=29, 63 | 0 | 3
  Total Bilirubin, G2, n=29, 63 | 0 | 0
  Total Bilirubin, G3, n=29, 63 | 0 | 0
  Total Bilirubin, G4, n=29, 63 | 0 | 0
  Albumin, G0, n=29, 63 | 29 | 63
  Albumin, G1, n=29, 63 | 0 | 0
  Albumin, G2, n=29, 63 | 0 | 0
  Albumin, G3, n=29, 63 | 0 | 0
  Albumin, G4, n=29, 63 | 0 | 0
  ALP, G0, n=29, 63 | 28 | 47
  ALP, G1, n=29, 63 | 1 | 16
  ALP, G2, n=29, 63 | 0 | 0
  ALP, G3, n=29, 63 | 0 | 0
  ALP, G4, n=29, 63 | 0 | 0
  PT INR, G0, n=27, 58 | 26 | 57
  PT INR, G1, n=27, 58 | 1 | 1
  PT INR, G2, n=27, 58 | 0 | 0
  PT INR, G3, n=27, 58 | 0 | 0
  PT INR, G4, n=27, 58 | 0 | 0
  APTT, G0 n=27, 58 | 13 | 24
  APTT, G1, n=27, 58 | 13 | 32
  APTT, G2, n=27, 58 | 1 | 2
  APTT, G3, n=27, 58 | 0 | 0
  APTT, G4, n=27, 58 | 0 | 0
  Creatinine, G0, n=29, 63 | 22 | 47
  Creatinine, G1, n=29, 63 | 7 | 15
  Creatinine, G2, n=29, 63 | 0 | 1
  Creatinine, G3, n=29, 63 | 0 | 0
  Creatinine, G4, n=29, 63 | 0 | 0

18. Secondary Outcome: Number of Participants With the Indicated Maximum Toxicity Grade for the Indicated Clinical Chemistry Parameters at Any Time Post-Baseline During Part 2
Description: Clinical chemistry parameters were summarized according to the NCI CTCAE, version 4.0: G0, none; G1, mild; G2, moderate; G3, severe; G4, life-threatening or disabling. Clinical chemistry parameters included: AST, ALP, total bilirubin, albumin, ALT, and creatinine. For participants randomized to Placebo in Part 1, the BL value for Part 2 is defined as the value taken at Week 13 of Part 1. For serum creatinine, the value taken at Week 13 of Part 1 will be used as BL. For participants randomized to Eltrombopag in Part 1, the BL value is defined as the value taken on Day 1 or, if missing, the latest non-missing Screening value. For serum creatinine, due to the variations in creatinine, the average of the Screening and the Day 1 values will be used as BL. For participants who do not have both a Screening and Day 1 value, the Screening or Day 1 value will be used as BL. The maximum post-BL toxicity grade includes any scheduled or unscheduled post-BL assessment.
Time Frame: From Baseline (BL) of Part 2 through Follow-up
Population: Safety Population. Only those participants who entered into Part 2 (Open-label eltrombopag-only phase) were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 2 (Open-Label Period) - Eltrombopag
Number analyzed (Participants) | 87
Participants
  AST, G0 | 63
  AST, G1 | 21
  AST, G2 | 1
  AST, G3 | 2
  AST, G4 | 0
  ALT, G0 | 67
  ALT, G1 | 14
  ALT, G2 | 3
  ALT, G3 | 3
  ALT, G4 | 0
  Total Bilirubin, G0 | 80
  Total Bilirubin, G1 | 4
  Total Bilirubin, G2 | 3
  Total Bilirubin, G3 | 0
  Total Bilirubin, G4 | 0
  Albumin, G0 | 85
  Albumin, G1 | 1
  Albumin, G2 | 1
  Albumin, G3 | 0
  Albumin, G4 | 0
  ALP, G0 | 67
  ALP, G1 | 20
  ALP, G2 | 0
  ALP, G3 | 0
  ALP, G4 | 0
  Creatinine, G0 | 72
  Creatinine, G1 | 14
  Creatinine, G2 | 1
  Creatinine, G3 | 0
  Creatinine, G4 | 0

19. Secondary Outcome: Number of Participants With the Indicated Maximum Toxicity Grade for the Indicated Hematology Parameters at Any Time Post-Baseline During Part 1
Description: Hematology parameters were summarized according to the NCI CTCAE, version 4.0: G0, none; G1, mild; G2, moderate; G3, severe; G4, life-threatening or disabling. Hematology parameters included: leukocytes, neutrophils, hemoglobin (increased), hemoglobin (anemia), lymphocytes (increased), and lymphocytes (decreased). The Baseline value is defined as the value taken at Day 1 or, if missing, the latest non-missing Screening value. The maximum post-Baseline toxicity grade includes any scheduled or unscheduled post-Baseline assessment during Part 1.
Time Frame: From Baseline up to Week 13 of Part 1
Population: as for outcome 17
Measure: Number; unit: Participants
Groups:
- Part 1(Randomized Period)-Placebo: In Part 1, participants aged between 6 and 17 years with a body weight <27 kg received placebo 37.5 mg QD, and those with a body weight >=27 kg received placebo 50 mg QD. Participants of East Asian ancestry received a starting dose of placebo 25 mg QD. Participants aged between 1 and 5 years received placebo 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of placebo 0.8 mg/kg/day.
Arm/Group | Part 1(Randomized Period)-Placebo | Part 1 (Randomized Period) - Eltrombopag
Number analyzed (Participants) | 29 | 63
Participants
  Leukocytes, G0, n=29, 63 | 23 | 50
  Leukocytes, G1, n=29, 63 | 6 | 11
  Leukocytes, G2, n=29, 63 | 0 | 0
  Leukocytes, G3, n=29, 63 | 0 | 1
  Leukocytes, G4, n=29, 63 | 0 | 1
  Neutrophils G0, n=29, 63 | 27 | 52
  Neutrophils G1, n=29, 63 | 1 | 3
  Neutrophils G2, n=29, 63 | 0 | 6
  Neutrophils G3, n=29, 63 | 1 | 0
  Neutrophils G4, n=29, 63 | 0 | 2
  Hemoglobin (increased), G0, n=29, 63 | 26 | 49
  Hemoglobin (increased), G1, n=29, 63 | 3 | 12
  Hemoglobin (increased), G2, n=29, 63 | 0 | 2
  Hemoglobin (increased), G3, n=29, 63 | 0 | 0
  Hemoglobin (increased), G4, n=29, 63 | 0 | 0
  Hemoglobin (anemia), G0, n=29, 63 | 20 | 42
  Hemoglobin (anemia), G1, n=29, 63 | 7 | 17
  Hemoglobin (anemia), G2, n=29, 63 | 0 | 4
  Hemoglobin (anemia), G3, n=29, 63 | 2 | 0
  Hemoglobin (anemia), G4, n=29, 63 | 0 | 0
  Lymphocytes (increased), G0, n=29, 63 | 17 | 37
  Lymphocytes (increased), G1, n=29, 63 | 0 | 0
  Lymphocytes (increased), G2, n=29, 63 | 12 | 26
  Lymphocytes (increased), G3, n=29, 63 | 0 | 0
  Lymphocytes (increased), G4, n=29, 63 | 0 | 0
  Lymphocytes (decreased), G0, n=29, 63 | 25 | 48
  Lymphocytes (decreased), G1, n=29, 63 | 4 | 13
  Lymphocytes (decreased), G2, n=29, 63 | 0 | 1
  Lymphocytes (decreased), G3, n=29, 63 | 0 | 1
  Lymphocytes (decreased), G4, n=29, 63 | 0 | 0

20. Secondary Outcome: Number of Participants With the Indicated Maximum Toxicity Grade for the Indicated Hematology Parameters at Any Time Post-Baseline During Part 2
Description: Hematology parameters were summarized according to the NCI CTCAE, version 4.0: G0, none, G1, mild; G2, moderate; G3, severe; G4, life-threatening or disabling. Hematology parameters included: leukocytes, neutrophils, hemoglobin (increased), hemoglobin (anemia), lymphocytes (increased), and lymphocytes (decreased). For participants randomized to Placebo in Part 1, the BL value for Part 2 is defined as the value taken at Week 13 of Part 1. For participants randomized to Eltrombopag in Part 1, the BL value is defined as the value taken on Day 1 or, if missing, the latest non-missing Screening value. For participants who do not have both a Screening and Day 1 value, the Screening or Day 1 value will be used as BL. The maximum post-BL toxicity grade includes any scheduled or unscheduled post-BL assessment.
Time Frame: From Baseline up to Week 24 of Part 2 and Follow-up Weeks 1 to 4 (up to Study Week 41)
Population: Safety Population. Only those participants who entered into Part 2 (Open-label eltrombopag-only phase) were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 2 (Open-Label Period) - Eltrombopag
Number analyzed (Participants) | 87
Participants
  Leukocytes, G0 | 59
  Leukocytes, G1 | 23
  Leukocytes, G2 | 3
  Leukocytes, G3 | 2
  Leukocytes, G4 | 0
  Neutrophils, G0 | 63
  Neutrophils, G1 | 6
  Neutrophils, G2 | 13
  Neutrophils, G3 | 2
  Neutrophils, G4 | 3
  Hemoglobin (increased), G0 | 74
  Hemoglobin (increased), G1 | 11
  Hemoglobin (increased), G2 | 2
  Hemoglobin (increased), G3 | 0
  Hemoglobin (increased), G4 | 0
  Hemoglobin (anemia), G0 | 48
  Hemoglobin (anemia), G1 | 31
  Hemoglobin (anemia), G2 | 7
  Hemoglobin (anemia), G3 | 1
  Hemoglobin (anemia), G4 | 0
  Lymphocytes (increased), G0 | 47
  Lymphocytes (increased), G1 | 0
  Lymphocytes (increased), G2 | 40
  Lymphocytes (increased), G3 | 0
  Lymphocytes (increased), G4 | 0
  Lymphocytes (decreased), G0 | 65
  Lymphocytes (decreased), G1 | 19
  Lymphocytes (decreased), G2 | 2
  Lymphocytes (decreased), G3 | 1
  Lymphocytes (decreased), G4 | 0

21. Secondary Outcome: Number of Participants With Vital Sign Data Falling Outside the Reference Ranges (RR) at the Indicated Visit During Part 1
Description: Vital sign measurements were taken before any blood draws and included systolic blood pressure(SBP), diastolic blood pressure(DBP), and heart rate(HR). The number of participants are reported with vital sign data falling outside the standard reference ranges RR as reference range high(RRH) and reference range low(RRL). The Baseline(BL) value is defined as the value taken at Day 1 or if missing, the latest non-missing SCR value. RR for Blood Pressure (mmHg) are read as: Lower Limit of Normal, Normal Range, Upper Limit of Normal. For Ages 1 to 5 years (yrs) ranges are SBP <85, 85 to 115, >115; DBP <45, 45 to70, >70. Ages 6 to 11 yrs: SBP <85, 85 to 120, >120;, DBP <50, 50 to 75, >75. Ages 12 to 17 yrs: SBP <95, 95 to 135, >135; DBP <55, 55 to 85, >85. RR for HR(bpm) are ages 1 to < 3 yrs: <90, 90 to 140, >140; ages 3 to < 5 yrs: <75, 75 to 130, >130, ages 5 to < 8yrs: <65, 65 to 115, >115; ages 8 to < 12yrs: <55, 55 to 110, >110; and ages 12 to 18 yrs: <55, 55 to 110, >110.
Time Frame: From Screening (SCR) up to Week 13 of Part 1
Population: as for outcome 17
Measure: Number; unit: Participants
Arm/Group | Part 1 (Randomized Period)-Placebo | Part 1 (Randomized Period)-Eltrombopag
Number analyzed (Participants) | 29 | 63
Participants
  DBP, Day 1, RRH, n=28,62 | 6 | 8
  DBP, Day 1, RRL, n=28, 62 | 2 | 5
  DBP, Week 1, RRH, n=28, 63 | 3 | 10
  DBP, Week 1, RRL, n=28, 63 | 0 | 5
  DBP, Week 2, RRH, n=29, 63 | 3 | 8
  DBP, Week 2, RRL, n=29, 63 | 2 | 6
  DBP, Week 3, RRH, n=28, 63 | 7 | 12
  DBP, Week 3, RRL, n=28, 63 | 2 | 6
  DBP, Week 4, RRH, n=29, 62 | 7 | 5
  DBP, Week 4, RRL, n=29, 62 | 2 | 9
  DBP, Week 5, RRH, n=27, 62 | 4 | 10
  DBP, Week 5, RRL, n=27, 62 | 2 | 6
  DBP, Week 6, RRH, n=28, 62 | 7 | 10
  DBP, Week 6, RRL, n=28, 62 | 1 | 8
  DBP, Week 7, RRH, n=28, 63 | 3 | 7
  DBP, Week 7, RRL, n=28, 63 | 2 | 5
  DBP, Week 8, RRH, n=28, 63 | 4 | 9
  DBP, Week 8, RRL, n=28, 63 | 2 | 8
  DBP, Week 9, RRH, n=27, 61 | 4 | 9
  DBP, Week 9, RRL, n=27, 61 | 2 | 4
  DBP, Week 10, RRH, n=28, 62 | 6 | 8
  DBP, Week 10, RRL, n=28, 62 | 2 | 7
  DBP, Week 11, RRH, n=28, 61 | 6 | 8
  DBP, Week 11, RRL, n=28, 61 | 3 | 6
  DBP, Week 12, RRH, n=28, 61 | 3 | 8
  DBP, Week 12, RRL, n=28, 61 | 0 | 6
  DBP, Week 13, RRH, n=28, 61 | 4 | 9
  DBP, Week 13, RRL, n=28, 61 | 3 | 4
  Heart Rate, Day 1, RRH, n=28, 62 | 0 | 2
  Heart Rate, Day 1, RRL, n=28, 62 | 0 | 1
  Heart Rate, Week 1, RRH, n=28, 63 | 0 | 0
  Heart Rate, Week 1, RRL, n=28, 63 | 0 | 0
  Heart Rate, Week 2, RRH, n=29, 63 | 2 | 1
  Heart Rate, Week 2, RRL, n=29, 63 | 0 | 1
  Heart Rate, Week 3, RRH, n=28, 63 | 1 | 2
  Heart Rate, Week 3, RRL, n=28, 63 | 0 | 0
  Heart Rate, Week 4, RRH, n=29, 61 | 0 | 4
  Heart Rate, Week 4, RRL, n=29, 61 | 0 | 1
  Heart Rate, Week 5, RRH, n=27, 62 | 1 | 5
  Heart Rate, Week 5, RRL, n=27, 62 | 1 | 0
  Heart Rate, Week 6, RRH, n=28,62 | 1 | 1
  Heart Rate, Week 6, RRL, n=28, 62 | 1 | 0
  Heart Rate, Week 7, RRH, n=28, 63 | 0 | 2
  Heart Rate, Week 7, RRL, n=28, 63 | 1 | 0
  Heart Rate, Week 8, RRH, n=28, 63 | 1 | 2
  Heart Rate, Week 8, RRL, n=28, 63 | 1 | 0
  Heart Rate, Week 9, RRH, n=27, 61 | 1 | 2
  Heart Rate, Week 9, RRL, n=27, 61 | 0 | 0
  Heart Rate, Week 10, RRH, n=28, 62 | 1 | 1
  Heart Rate, Week 10, RRL, n=28, 62 | 0 | 0
  Heart Rate, Week 11, RRH, n=28, 61 | 1 | 2
  Heart Rate, Week 11, RRL, n=28, 61 | 0 | 0
  Heart Rate, Week 12, RRH, n=28,61 | 0 | 2
  Heart Rate, Week 12, RRL, n=28, 61 | 0 | 0
  Heart Rate, Week 13, RRH, n=28, 61 | 0 | 3
  Heart Rate, Week 13, RRL, n=28, 61 | 1 | 0
  SBP, Day 1, RRH, n=28, 62 | 5 | 10
  SBP, Day 1, RRL, n=28, 62 | 3 | 6
  SBP, Week 1, RRH, n=28, 63 | 3 | 11
  SBP, Week 1, RRL, n=28,63 | 4 | 8
  SBP, Week 2, RRH, n=29, 63 | 4 | 7
  SBP, Week 2, RRL, n=29, 63 | 3 | 9
  SBP, Week 3, RRH, n=28, 63 | 3 | 9
  SBP, Week 3, RRL, n=28, 63 | 2 | 9
  SBP, Week 4, RRH, n=29, 62 | 3 | 10
  SBP, Week 4, RRL, n=29, 62 | 2 | 9
  SBP, Week 5, RRH, n=27, 62 | 5 | 9
  SBP, Week 5, RRL, n=27, 62 | 4 | 7
  SBP, Week 6, RRH, n=28, 62 | 5 | 7
  SBP, Week 6, RRL, n=28, 62 | 3 | 8
  SBP, Week 7, RRH, n=28, 63 | 5 | 10
  SBP, Week 7, RRL, n=28, 63 | 3 | 7
  SBP, Week 8, RRH, n=28, 63 | 3 | 14
  SBP, Week 8, RRL, n=28, 63 | 4 | 7
  SBP, Week 9, RRH, n=27, 61 | 4 | 12
  SBP, Week 9, RRL, n=27, 61 | 3 | 7
  SBP, Week 10, RRH, n=28, 62 | 4 | 11
  SBP, Week 10, RRL, n=28, 62 | 3 | 11
  SBP, Week 11, RRH, n=28, 61 | 6 | 12
  SBP, Week 11, RRL, n=28, 61 | 5 | 9
  SBP, Week 12, RRH, n=28, 61 | 4 | 11
  SBP, Week 12, RRL, n=28, 61 | 4 | 4
  SBP, Week 13, RRH, n=28, 61 | 6 | 9
  SBP, Week 13, RRL, n=28, 61 | 4 | 7

22. Secondary Outcome: Number of Participants With Vital Sign Data Falling Outside the Reference Ranges (RR) at the Indicated Visit During Part 2
Description: Vital sign measurements were taken before any blood draw and included systolic blood pressure (SBP), diastolic blood pressure (DBP), and heart rate(HR). The number of participants are reported with vital sign data falling outside the standard RR as reference range high(RRH) and reference range low(RRL) from SCR up to Week 24 of Part 2 and from Follow-up Week 1 to Week 4. RR for Blood Pressure(mmHg) are read as: Lower Limit of Normal, Normal Range, Upper Limit of Normal. For Ages 1 to 5 years (yrs) ranges are SBP <85, 85 to 115, >115; DBP <45, 45 to70, >70. Ages 6 to 11 yrs: SBP <85, 85 to 120, >120; DBP <50, 50 to 75, >75. Ages 12 to 17 yrs: SBP <95, 95 to 135, >135; DBP <55, 55 to 85, >85. RR for HR (bpm) are ages 1 to < 3 yrs: <90, 90 to 140, >140; ages 3 to < 5 yrs: <75, 75 to 130, >130, ages 5 to < 8yrs: <65, 65 to 115, >115; ages 8 to < 12yrs: <55, 55 to 110, >110; and ages 12 to 18 yrs: <55, 55 to 110, >110.
Time Frame: From Week 1 up to Week 24 of Part 2 and Follow-up Week 1 to Week 4 (up to Week 41)
Population: Safety Population. Only those participants who entered into Part 2 (Open-label eltrombopag-only phase) were analyzed. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Number; unit: Participants
Arm/Group | Part 2 (Open-Label Period) - Eltrombopag
Number analyzed (Participants) | 87
Participants
  DBP, Week 1, RRH, n=87 | 14
  DBP, Week 1, RRL, n=87 | 8
  DBP, Week 2, RRH, n=86 | 14
  DBP, Week 2, RRL, n=86 | 8
  DBP, Week 3, RRH, n=86 | 13
  DBP, Week 3, RRL, n=86 | 11
  DBP, Week 4, RRH, n=68 | 10
  DBP, Week 4, RRL, n=68 | 7
  DBP, Week 5, RRH, n=61 | 7
  DBP, Week 5, RRL, n=61 | 7
  DBP, Week 6, RRH, n=55 | 6
  DBP, Week 6, RRL, n=55 | 4
  DBP, Week 7, RRH, n=52 | 7
  DBP, Week 7, RRL, n=52 | 5
  DBP, Week 8, RRH, n=53 | 4
  DBP, Week 8, RRL, n=53 | 6
  DBP, Week 9, RRH, n=45 | 3
  DBP, Week 9, RRL, n=45 | 7
  DBP, Week 10, RRH, n=42 | 5
  DBP, Week 10, RRL, n=42 | 7
  DBP, Week 11, RRH, n=40 | 5
  DBP, Week 11, RRL, n=40 | 7
  DBP, Week 12, RRH, n=63 | 9
  DBP, Week 12, RRL, n=63 | 11
  DBP, Week 13, RRH, n=29 | 4
  DBP, Week 13, RRL, n=29 | 2
  DBP, Week 14, RRH, n=38 | 2
  DBP, Week 14, RRL, n=38 | 9
  DBP, Week 15, RRH, n=43 | 7
  DBP, Week 15, RRL, n=43 | 3
  DBP, Week 16, RRH, n=47 | 3
  DBP, Week 16, RRL, n=47 | 6
  DBP, Week 17, RRH, n=37 | 5
  DBP, Week 17, RRL, n=37 | 6
  DBP, Week 18, RRH, n=34 | 7
  DBP, Week 18, RRL, n=34 | 5
  DBP, Week 19, RRH, n=44 | 5
  DBP, Week 19, RRL, n=44 | 3
  DBP, Week 20, RRH, n=39 | 6
  DBP, Week 20, RRL, n=39 | 3
  DBP, Week 21, RRH, n=41 | 9
  DBP, Week 21, RRL, n=41 | 6
  DBP, Week 22, RRH, n=34 | 6
  DBP, Week 22, RRL, n=34 | 3
  DBP, Week 23, RRH, n=36 | 6
  DBP, Week 23, RRL, n=36 | 6
  DBP, Week 24, RRH, n=79 | 14
  DBP, Week 24, RRL, n=79 | 10
  DBP, Follow-Up Week 1, RRH, n=29 | 8
  DBP, Follow-Up Week 1, RRL, n=29 | 3
  DBP, Follow-Up Week 2, RRH, n=37 | 8
  DBP, Follow-Up Week 2, RRL, n=37 | 6
  DBP, Follow-Up Week 3, RRH, n=39 | 4
  DBP, Follow-Up Week 3, RRL, n=39 | 5
  DBP, Follow-Up Week 4, RRH, n=67 | 8
  DBP, Follow-Up Week 4, RRL, n=67 | 5
  Heart Rate, Week 1, RRH, n=87 | 4
  Heart Rate, Week 1, RRL, n=87 | 1
  Heart Rate, Week 2, RRH, n=86 | 3
  Heart Rate, Week 2, RRL, n=86 | 2
  Heart Rate, Week 3, RRH, n=86 | 1
  Heart Rate, Week 3, RRL, n=86 | 0
  Heart Rate, Week 4, RRH, n=68 | 2
  Heart Rate, Week 4, RRL, n=68 | 0
  Heart Rate, Week 5, RRH, n=61 | 0
  Heart Rate, Week 5, RRL, n=61 | 1
  Heart Rate, Week 6, RRH, n=55 | 1
  Heart Rate, Week 6, RRL, n=55 | 0
  Heart Rate, Week 7, RRH, n=52 | 2
  Heart Rate, Week 7, RRL, n=52 | 0
  Heart Rate, Week 8, RRH, n=53 | 2
  Heart Rate, Week 8, RRL, n=53 | 0
  Heart Rate, Week 9, RRH, n=45 | 2
  Heart Rate, Week 9, RRL, n=45 | 0
  Heart Rate, Week 10, RRH, n=42 | 1
  Heart Rate, Week 10, RRL, n=42 | 1
  Heart Rate, Week 11, RRH, n=40 | 1
  Heart Rate, Week 11, RRL, n=40 | 1
  Heart Rate, Week 12, RRH, n=63 | 1
  Heart Rate, Week 12, RRL, n=63 | 1
  Heart Rate, Week 13, RRH, n=29 | 2
  Heart Rate, Week 13, RRL, n=29 | 0
  Heart Rate, Week 14, RRH, n=38 | 2
  Heart Rate, Week 14, RRL, n=38 | 1
  Heart Rate, Week 15, RRH, n=43 | 0
  Heart Rate, Week 15, RRL, n=43 | 0
  Heart Rate, Week 16, RRH, n=47 | 2
  Heart Rate, Week 16, RRL, n=47 | 0
  Heart Rate, Week 17, RRH, n=37 | 2
  Heart Rate, Week 17, RRL, n=37 | 1
  Heart Rate, Week 18, RRH, n=34 | 0
  Heart Rate, Week 18, RRL, n=34 | 0
  Heart Rate, Week 19, RRH, n=44 | 0
  Heart Rate, Week 19, RRL, n=44 | 1
  Heart Rate, Week 20, RRH, n=39 | 2
  Heart Rate, Week 20, RRL, n=39 | 0
  Heart Rate, Week 21, RRH, n=41 | 0
  Heart Rate, Week 21, RRL, n=41 | 0
  Heart Rate, Week 22, RRH, n=34 | 2
  Heart Rate, Week 22, RRL, n=34 | 0
  Heart Rate, Week 23, RRH, n=36 | 0
  Heart Rate, Week 23, RRL, n=36 | 0
  Heart Rate, Week 24, RRH, n=79 | 1
  Heart Rate, Week 24, RRL, n=79 | 1
  Heart Rate, Follow-Up Week 1, RRH, n=29 | 1
  Heart Rate, Follow-Up Week 1, RRL, n=29 | 0
  Heart Rate, Follow-Up Week 2, RRH, n=37 | 2
  Heart Rate, Follow-Up Week 2, RRL, n=37 | 1
  Heart Rate, Follow-Up Week 3, RRH, n=39 | 2
  Heart Rate, Follow-Up Week 3, RRL, n=39 | 0
  Heart Rate, Follow-Up Week 4, RRH, n=67 | 2
  Heart Rate, Follow-Up Week 4, RRL, n=67 | 2
  SBP, Week 1, RRH, n=87 | 13
  SBP, Week 1, RRL, n=87 | 9
  SBP, Week 2, RRH, n=86 | 19
  SBP, Week 2, RRL, n=86 | 16
  SBP, Week 3, RRH, n=86 | 15
  SBP, Week 3, RRL, n=86 | 13
  SBP, Week 4, RRH, n=68 | 10
  SBP, Week 4, RRL, n=68 | 7
  SBP, Week 5, RRH, n=61 | 7
  SBP, Week 5, RRL, n=61 | 8
  SBP, Week 6, RRH, n=55 | 11
  SBP, Week 6, RRL, n=55 | 7
  SBP, Week 7, RRH, n=52 | 10
  SBP, Week 7, RRL, n=52 | 5
  SBP, Week 8, RRH, n=53 | 8
  SBP, Week 8, RRL, n=53 | 5
  SBP, Week 9, RRH, n=45 | 8
  SBP, Week 9, RRL, n=45 | 9
  SBP, Week 10, RRH, n=42 | 4
  SBP, Week 10, RRL, n=42 | 4
  SBP, Week 11, RRH, n=40 | 4
  SBP, Week 11, RRL, n=40 | 6
  SBP, Week 12, RRH, n=63 | 14
  SBP, Week 12, RRL, n=63 | 10
  SBP, Week 13, RRH, n=29 | 3
  SBP, Week 13, RRL, n=29 | 2
  SBP, Week 14, RRH, n=38 | 5
  SBP, Week 14, RRL, n=38 | 7
  SBP, Week 15, RRH, n=43 | 9
  SBP, Week 15, RRL, n=43 | 7
  SBP, Week 16, RRH, n=47 | 7
  SBP, Week 16, RRL, n=47 | 6
  SBP, Week 17, RRH, n=37 | 9
  SBP, Week 17, RRL, n=37 | 4
  SBP, Week 18, RRH, n=34 | 6
  SBP, Week 18, RRL, n=34 | 5
  SBP, Week 19, RRH, n=44 | 7
  SBP, Week 19, RRL, n=44 | 4
  SBP, Week 20, RRH, n=39 | 5
  SBP, Week 20, RRL, n=39 | 5
  SBP, Week 21, RRH, n=41 | 10
  SBP, Week 21, RRL, n=41 | 6
  SBP, Week 22, RRH, n=34 | 6
  SBP, Week 22, RRL, n=34 | 4
  SBP, Week 23, RRH, n=36 | 6
  SBP, Week 23, RRL, n=36 | 3
  SBP, Week 24, RRH, n=79 | 13
  SBP, Week 24, RRL, n=79 | 12
  SBP, Follow-Up Week 1, RRH, n=29 | 5
  SBP, Follow-Up Week 1, RRL, n=29 | 3
  SBP, Follow-Up Week 2, RRH, n=37 | 5
  SBP, Follow-Up Week 2, RRL, n=37 | 7
  SBP, Follow-Up Week 3, RRH, n=39 | 9
  SBP, Follow-Up Week 3, RRL, n=39 | 4
  SBP, Follow-Up Week 4, RRH, n=67 | 9
  SBP, Follow-Up Week 4, RRL, n=67 | 7

23. Secondary Outcome: Number of Participants With a Change in Visual Acuity Since Baseline at Week 12 of Part 1
Description: The visual acuity assessment was performed by an ophthalmologist or an optometrist under the guidance of an ophthalmologist. Visual acuity is defined as acuteness or clearness of vision. Change in visual acuity results are presented as No (no change from Baseline), Not Clinically Significant (NCS), Improvement, and Worsening since Baseline. The Baseline value was obtained at the Screening Visit.
Time Frame: Baseline and Week 12 of Part 1
Population: Safety Population
Measure: Number; unit: Participants
Groups:
- EPart 1 (Randomized Period)-Placebo: In Part 1, participants aged between 6 and 17 years with a body weight <27 kg received placebo 37.5 mg QD, and those with a body weight >=27 kg received placebo 50 mg QD. Participants of East Asian ancestry received a starting dose of placebo 25 mg QD. Participants aged between 1 and 5 years received placebo 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of placebo 0.8 mg/kg/day.
Arm/Group | EPart 1 (Randomized Period)-Placebo | Part 1 (Randomized Period)-Eltrombopag
Number analyzed (Participants) | 29 | 63
Participants
  No Change | 22 | 47
  NCS | 4 | 8
  Improvement | 1 | 2
  Worsening | 0 | 1
  Not Measured | 2 | 5

24. Secondary Outcome: Number of Participants With a Change in Visual Acuity Since Baseline at Week 24 of Part 2
Description: The visual acuity assessment was performed by an ophthalmologist or an optometrist under the guidance of an ophthalmologist. Visual acuity is defined as acuteness or clearness of vision. Change in visual acuity results are presented as No Change, NCS, Improvement, and Worsening since Baseline. The Baseline value was obtained at the Screening Visit.
Time Frame: Baseline and Week 24 of Part 2
Population: Safety Population. Only those participants who entered into Part 2 (Open-label eltrombopag-only phase) were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 2 (Open-Label Period) - Eltrombopag
Number analyzed (Participants) | 87
Participants
  No Change | 58
  NCS | 13
  Improvement | 3
  Worsening | 6
  Not Measured | 7

25. Secondary Outcome: Number of Participants With a Change in Visual Acuity Since Baseline at Follow-Up Week 24
Description: as for outcome 24
Time Frame: Baseline and Follow-Up Week 24 (Study Week 61)
Population: Safety Population. Only those participants who entered into Part 2 (Open-label eltrombopag-only phase) were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 2 (Open-Label Period) - Eltrombopag
Number analyzed (Participants) | 87
Participants
  No Change | 63
  NCS | 12
  Improvement | 9
  Worsening | 2
  Not Measured | 1

26. Secondary Outcome: Number of Participants With Worsening Visual Acuity Due to Cataracts at Week 12 of Part 1
Description: The visual acuity assessment was performed by an ophthalmologist or an optometrist under the guidance of an ophthalmologist. Visual acuity is defined as acuteness or clearness of vision. The number of participants with worsening visual acuity due to cataracts at Week 12 of Part 1 are presented. Change due to cataracts is categorized as "Yes" or "No."
Time Frame: Baseline and Week 12 of Part 1
Population: Safety Population. Only those participants who had a result of 'worsening' in assessment of change of visual acuity at this timepoint were analyzed.
Measure: Number; unit: Participants
Groups:
- Part 1 (Randomized Period) - Placebo: In Part 1, participants aged between 6 and 17 years with a body weight <27 kg received placebo 37.5 mg QD, and those with a body weight >=27 kg received placebo 50 mg QD. Participants of East Asian ancestry received a starting dose of placebo 25 mg QD. Participants aged between 1 and 5 years received placebo 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of placebo 0.8 mg/kg/day.
Arm/Group | Part 1 (Randomized Period) - Placebo | Part 1 (Randomized Period) - Eltrombopag
Number analyzed (Participants) | 0 | 1
Participants
  Yes |  | 0
  No |  | 1

27. Secondary Outcome: Number of Participants With Worsening Visual Acuity Due to Cataracts at Week 24 of Part 2
Description: The visual acuity assessment was performed by an ophthalmologist or an optometrist under the guidance of an ophthalmologist. Visual acuity is defined as acuteness or clearness of vision. The number of participants with worsening visual acuity due to cataracts at Week 24 of Part 2 are presented. Change due to cataracts is categorized as "Yes" or "No.
Time Frame: Baseline and Week 24 of Part 2
Population: Safety Population. Only those participants who had worsening visual acuity at Week 24 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 2 (Open-Label Period) - Eltrombopag
Number analyzed (Participants) | 6
Participants
  Yes | 1
  No | 5

28. Secondary Outcome: Number of Participants With Worsening Visual Acuity Due to Cataracts at Follow-Up Week 24
Description: The visual acuity assessment was performed by an ophthalmologist or an optometrist under the guidance of an ophthalmologist. Visual acuity is defined as acuteness or clearness of vision. The number of participants with worsening visual acuity due to cataracts at Follow-up Week 24 are presented. Change due to cataracts is categorized as "Yes" or "No."
Time Frame: Baseline and Follow-Up Week 24 (Week 61)
Population: Safety Population. Only those participants who had worsening visual acuity at Week 61 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Part 2 (Open-Label Period) - Eltrombopag
Number analyzed (Participants) | 2
Participants
  Yes | 0
  No | 2

29. Secondary Outcome: Pharmacokinetic (PK) Assessments for Eltrombopag for AUC (0-t)
Description: Single PK samples were collected at each visit during Part 1 Weeks 2, 4, 6, 8, 10, 12 and at each weekly or monthly visit during Part 2 Weeks 1-12 (Study Weeks 13-37). The concentration data were pooled across visits to identify population PK and variability parameter estimates and covariate effects. AUC(0-t) is defined as the area under the concentration-time curve over the dosing interval. The AUC(0-t) for a 50mg dose was estimated for each cohort. From the final model, a single value of each PK parameter was estimated for each subject, and geometric mean (95% CI) values are presented for each cohort for a 50mg dose.
Time Frame: Part 1 Weeks 2, 4, 6, 8, 10, 12, and Part 2 Weeks 1-12 (Study Weeks 13 - 37)
Population: PK Population. Only those participants who provided pharmacokinetic samples were analyzed
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms*hour per milliliter (ug.h/mL)
Groups:
- Eltrombopag Cohort 1 (12-17 Years): Participants who received eltrombopag in Part 1 continued on the same dose in Part 2 unless adjustments were warranted according to the dosing guidelines. Participants who received placebo in Part 1 received Eltrombopag as per age criteria as follows:body weight <27 kg received eltrombopag 37.5 mg QD, and those with a body weight >=27 kg received eltrombopag 50 mg QD. Participants of East Asian ancestry received a starting dose of eltrombopag 25 mg QD.
- Eltrombopag Cohort 2 (6-11 Years): Participants who received eltrombopag in Part 1 continued on the same dose in Part 2 unless adjustments were warranted according to the dosing guidelines. Participants who received placebo in Part 1 received Eltrombopag as per age criteria as follows: body weight <27 kg received eltrombopag 37.5 mg QD, and those with a body weight >=27 kg received eltrombopag 50 mg QD. Participants of East Asian ancestry received a starting dose of eltrombopag 25 mg QD.
- Eltrombopag Cohort 3 (1-5 Years): Participants who received eltrombopag in Part 1 continued on the same dose in Part 2 unless adjustments were warranted according to the dosing guidelines. Participants who received placebo in Part 1 received Eltrombopag 1.2 mg/kg QD and; participants of East Asian ancestry received a starting dose of eltrombopag 0.8 mg/kg/day.
Arm/Group | Eltrombopag Cohort 1 (12-17 Years) | Eltrombopag Cohort 2 (6-11 Years) | Eltrombopag Cohort 3 (1-5 Years)
Number analyzed (Participants) | 33 | 38 | 19
micrograms*hour per milliliter (ug.h/mL) | 104 [86.1 to 126] | 171 [147 to 200] | 184 [147 to 230]

30. Secondary Outcome: Pharmacokinetic (PK) Assessments for Eltrombopag for Cmax
Description: Single PK samples were collected at each visit during Part 1 Weeks 2, 4, 6, 8, 10, 12 and at each weekly or monthly visit during Part 2 Weeks 1-12 (Study Weeks 13-37). The concentration data were pooled across visits to identify population PK and variability parameter estimates and covariate effects. Cmax is defined as the maximum observed concentration. The Cmax for a 50mg dose was estimated for each cohort. From the final model, a single value of each PK parameter was estimated for each subject, and geometric mean (95% CI) values are presented for each cohort for a 50mg dose.
Time Frame: Part 1 Weeks 2, 4, 6, 8, 10, 12, and Part 2 Weeks 1-12 (Study Weeks 13 - 37)
Population: PK Population. Only those participants who provided pharmacokinetic samples were analyzed
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms per milliliter (ug/mL)
Arm/Group | Eltrombopag Cohort 1 (12-17 Years) | Eltrombopag Cohort 2 (6-11 Years) | Eltrombopag Cohort 3 (1-5 Years)
Number analyzed (Participants) | 33 | 38 | 19
micrograms per milliliter (ug/mL) | 6.94 [5.96 to 8.08] | 11.2 [9.91 to 12.8] | 12.5 [10.7 to 14.6]

31. Secondary Outcome: Pharmacokinetic (PK) Assessments for Eltrombopag for Apparent Oral Clearance (CL/F) and Apparent Intercompartmental Clearance (Q/F)
Description: Single PK samples were collected at each visit during Part 1 Weeks 2, 4, 6, 8, 10, 12 and at each weekly or monthly visit during Part 2 Weeks 1-12 (Study Weeks 13-37). The concentration data were pooled across visits to identify population PK and variability parameter estimates and covariate effects. CL/F is defined as the apparent oral clearance from plasma and Q/F is defined as apparent intercompartmental clearance. These parameters are dose independent. From the final model, a single value of each PK parameter was estimated for each subject, and geometric mean (95% CI) values are presented for each cohort.
Time Frame: Part 1 Weeks 2, 4, 6, 8, 10, 12, and Part 2 Weeks 1-12 (Study Weeks 13 - 37)
Population: PK Population. Only those participants who provided pharmacokinetic samples were analyzed
Measure: Geometric Mean (95% Confidence Interval); unit: Liters per hour (L/hr)
Arm/Group | Eltrombopag Cohort 1 (12-17 Years) | Eltrombopag Cohort 2 (6-11 Years) | Eltrombopag Cohort 3 (1-5 Years)
Number analyzed (Participants) | 33 | 38 | 19
Liters per hour (L/hr)
  CL/F | 0.48 [0.40 to 0.58] | 0.29 [0.25 to 0.34] | 0.19 [0.15 to 0.24]
  Q/F | 0.61 [0.54 to 0.68] | 0.38 [0.34 to 0.42] | 0.24 [0.20 to 0.28]

32. Secondary Outcome: PK Assessments for Eltrombopag for Apparent Central Volume (Vc/F) and Apparent Peripheral Volume (Vp/F)
Description: Single PK samples were collected at each visit during Part 1 Weeks 2, 4, 6, 8, 10, 12 and at each weekly or monthly visit during Part 2 Weeks 1-12 (Study Weeks 13-37). The concentration data were pooled across visits to identify population PK and variability parameter estimates and covariate effects. Vc/F is defined as the volume of the central (e.g. plasma) compartment and Vp/F is defined as the volume of the peripheral compartment. These parameters are dose independent. From the final model, a single value of each PK parameter was estimated for each subject, and geometric mean (95% CI) values are presented for each cohort.
Time Frame: Part 1 Weeks 2, 4, 6, 8, 10, 12, and Part 2 Weeks 1-12 (Study Weeks 13 - 37)
Population: PK Population. Only those participants who provided pharmacokinetic samples were analyzed
Measure: Geometric Mean (95% Confidence Interval); unit: Liters (L)
Arm/Group | Eltrombopag Cohort 1 (12-17 Years) | Eltrombopag Cohort 2 (6-11 Years) | Eltrombopag Cohort 3 (1-5 Years)
Number analyzed (Participants) | 33 | 38 | 19
Liters (L)
  Vc/F | 2.46 [2.20 to 2.75] | 1.57 [1.35 to 1.81] | 0.90 [0.76 to 1.05]
  Vp/F | 19.2 [17.7 to 20.9] | 11.8 [10.9 to 12.9] | 7.17 [6.58 to 7.81]

33. Secondary Outcome: Population PK Model Point Estimate for Eltrombopag for Absorption Rate-constant (Ka)
Description: Single PK samples were collected at each visit during Part 1 Weeks 2, 4, 6, 8, 10, 12 and at each weekly or monthly visit during Part 2 Weeks 1-12 (Study Weeks 13-37). The concentration data were pooled across visits to identify population PK and variability parameter estimates and covariate effects. Ka is defined as the absorption rate constant. This parameter is dose independent, and the population estimate Ka is reported.
Time Frame: Part 1 Weeks 2, 4, 6, 8, 10, 12, and Part 2 Weeks 1-12 (Study Weeks 13 - 37)
Population: PK Population. Only those participants who provided pharmacokinetic samples were analyzed
Measure: Number; unit: 1/h
Arm/Group | Eltrombopag Cohort 1 (12-17 Years) | Eltrombopag Cohort 2 (6-11 Years) | Eltrombopag Cohort 3 (1-5 Years)
Number analyzed (Participants) | 33 | 38 | 19
1/h | 0.189 | 0.189 | 0.189

ADVERSE EVENTS:
Time Frame: On-treatment adverse events (AEs) and serious adverse events (SAEs) are defined as events occuring from the start of investigational product until follow up (up to 61 weeks).
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all participants who had received at least one dose of the investigational product.
Groups:
- Part 1: Eltrombopag: In Part 1, participants aged between 6 and 17 years with a body weight less than 27 kg received eltrombopag 37.5 mg QD, and those with a body weight greater than or equal to 27 kg received eltrombopag 50 mg QD. Participants of East Asian ancestry received a starting dose of eltrombopag 25 mg QD. Participants aged between 1 and 5 years received eltrombopag 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of eltrombopag 0.8 mg/kg/day.
- Part 1: Placebo: In Part 1, participants aged between 6 and 17 years with a body weight less than 27 kg received placebo 37.5 mg QD, and those with a body weight greater than or equal to 27 kg received placebo 50 mg QD. Participants of East Asian ancestry received a starting dose of placebo 25 mg QD. Participants aged between 1 and 5 years received placebo 1.2 mg/kg QD; participants of East Asian ancestry received a starting dose of placebo 0.8 mg/kg/day.
- Part 2: Eltrombopag: In Part 2, participants continued on the same dose of eltrombopag received in Part 1 unless adjustments were warranted according to the dosing guidelines.
Arm/Group | Part 1: Eltrombopag | Part 1: Placebo | Part 2: Eltrombopag
Serious Adverse Events (participants affected / at risk) | 5/63 | 4/29 | 9/87
Other Adverse Events (participants affected / at risk) | 51/63 | 19/29 | 68/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Eltrombopag (N=63) | Part 1: Placebo (N=29) | Part 2: Eltrombopag (N=87)
Gingivitis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0
Alanine aminotransferase abnormal (Investigations) | 1 | 0 | 0
Aspartate aminotransferase abnormal (Investigations) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Eltrombopag (N=63) | Part 1: Placebo (N=29) | Part 2: Eltrombopag (N=87)
Nasopharyngitis (Infections and infestations) | 11 | 2 | 7
Rhinitis (Infections and infestations) | 10 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 8
Upper respiratory tract infection (Infections and infestations) | 7 | 1 | 9
Abdominal pain (Gastrointestinal disorders) | 6 | 0 | 7
Headache (Nervous system disorders) | 6 | 3 | 8
Aspartate Aminotransferase increased (Investigations) | 4 | 0 | 7
Pyrexia (General disorders) | 4 | 1 | 9
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4 | 3
Alanine Aminotransferase increased (Investigations) | 3 | 0 | 6
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Toothache (Gastrointestinal disorders) | 3 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0 | 0
Blood alkaline Phosphatase increased (Investigations) | 2 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 1 | 1
Bronchitis (Investigations) | 2 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 3
Gingival bleeding (Gastrointestinal disorders) | 2 | 1 | 2
Mouth haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 3 | 6
Allergy to chemicals (Immune system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 4
Asthenia (General disorders) | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bulimia nervosa (Psychiatric disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 2
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 2
Gingivitis (Infections and infestations) | 1 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Impetigo (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 1
Influenza like illness (General disorders) | 1 | 1 | 5
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lice infestation (Infections and infestations) | 1 | 0 | 2
Lip haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 1 | 1
Motion sickness (Ear and labyrinth disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 7
Platelet count increased (Investigations) | 1 | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Retinal vascular disorder (Eye disorders) | 1 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0 | 0
Blood albumin increased (Investigations) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0
Helminthic infection (Infections and infestations) | 0 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Otosalpingitis (Ear and labyrinth disorders) | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pericoronitis (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Tongue biting (Nervous system disorders) | 0 | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 6
Hyperaemia (Vascular disorders) | 0 | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 3
Viral infection (Infections and infestations) | 0 | 0 | 3
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Acute tonsillitis (Infections and infestations) | 0 | 0 | 1
Adenoiditis (Infections and infestations) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1
Essential hypertension (Vascular disorders) | 0 | 0 | 1
Eyelid infection (Infections and infestations) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Glucose-6-phosphate dehydrogenase deficiency (Congenital, familial and genetic disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 0 | 1
Infection parasitic (Infections and infestations) | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Menarche (Social circumstances) | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1
Migraine with aura (Nervous system disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pupils unequal (Eye disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Serum ferritin decreased (Investigations) | 0 | 0 | 1
Tic (Psychiatric disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.